CLINICAL TRIAL: NCT01863862
Title: Organ Preservation in Elderly Patients With Rectal Cancer: a Prospective Observational Study
Brief Title: Organ Preservation in Elderly Patients With Rectal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGBRJG0113
Record Dates: First submitted 2013-05-14; First posted 2013-05-29 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Chemoradiation; Complete pathological response
MeSH Terms: conditions — Rectal Neoplasms; Pathologic Complete Response | interventions — Chemoradiotherapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clinical complete responders. (Experimental): Patients with complete clinical response obtained 8 weeks after chemoradiation or 10 weeks after short-course radiation.
  Interventions: Radiation: Radiochemotherapy or radiotherapy

INTERVENTIONS:
Radiation: Radiochemotherapy or radiotherapy — 50 Gy, 2 Gy per fraction with simultaneous 5-Fu and leucovorin or 5 x 5 Gy for patients unfit for chemotherapy.
  Patients with complete clinical response 8-10 weeks after radiotherapy will be closely observed and rescue surgery will be performed in a case of local recurrence.
  Patients with persistent tumour 8-10 weeks after radiotherapy will undergo transanal endoscopic microsurgery or total mesorectal excision. After transanal endosciopic microsurgery, patients with ypT0-1 disease and negative surgical margins will be closely observed and rescue total mesorectal excision will be performed in a case of local recurrence; those with ypT2-3 disease or with positive margin will undergo immediate conversion to total mesorectal excision.

SUMMARY:
In elderly patients postoperative mortality measured 3-6 months after total mesorectal excision is high. Thus, less toxic treatments may lead to a survival benefit for elderly patients even if a risk of local recurrence is slightly higher compared to the open surgery. The investigators addressed the question whether watch and wait policy is safe in clinical complete responders after (chemo)radiation for elderly patients with small or moderately advanced tumours.

DETAILED DESCRIPTION:
There are two steps of selection. In the first step, the elderly patients with small or moderately advanced tumours who should routinely receive neoadjuvant chemoradiation (or radiation alone in those unfit for chemotherapy) prior to full-thickness local excision using transanal endoscopic microsurgery or prior to total mesorectal excision will be included. In the next step, only patients with clinical complete response obtained 8-10 weeks from completion of (chemo)radiation are selected. Those patients constitute study group and will be observed without further treatment. The remaining patients with residual cancer will proceed to routine management, namely transanal endoscopic microsurgery or total mesorectal excision. Patients undergoing transanal endoscopic microsurgery and having poor response to (chemo)radiation (ypT2-3 disease or positive margin) will proceed to the conversion to total mesorectal excision.

Neoadjuvant chemoradiation: 50 Gy total dose over 5 weeks with 2 Gy per fraction delivered with simultaneous chemotherapy consisting of three cycles of 5-Fu 200 mg/m2 i.v. bolus and leucovorin 100 mg/m2 i.v. short infusion over 2 days given during 1-2, 15-16, and 29-30 days of radiotherapy. Patients unfit for chemotherapy will receive 25 Gy total dose over 5 days with 5 Gy per fraction.

The study hypothesis is that in clinical complete responders after (chemo)radiation treated without initial surgery, the local recurrence rate will be less than 25% and results of the rescue surgery (local and distant recurrence rate) will be not worse (or only slightly worse) than that seen after up-front total mesorectal excision in patients with similar stage of the disease.

ELIGIBILITY:
Inclusion Criteria:

The initial eligibility criteria

* Age ≥70 years or <70 years in patients with ASA 3+
* Tumour accessible by digital rectal examination
* Maximal tumour size (usually length) not more than 5 cm
* Circumferential bowel wall involvement not larger than 60%

There will be two groups of patients:

1. Candidates for preoperative (chemo)radiotherapy and local excision: tumour ≤3 cm, non-polipoid cT1, or cT2 or borderline cT3, cN0.
2. Candidates for preoperative (chemo)radiotherapy and total mesorectal excision: cT2 tumors requiring abdominoperineal excision, or cT3 or resectable cT4 (slight involvement of vagina, prostate or seminal vesicles); cN+ is allowed.

The final eligibility criterion

• Complete clinical response obtained 8 weeks after chemoradiation or 10 weeks after short-course radiation

Exclusion Criteria:

* Distant metastases
* Fixed tumour on digital rectal examination

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-08; Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
The final three-year rate of local and distant recurrences taking into consideration results of rescue surgery for pelvic recurrence. | After 3 years of median follow-up for living patients.

SECONDARY OUTCOMES:
The rate of local recurrence at one year without taking into consideration results of rescue surgery. | up to 20 months
The rate of local and distant recurrences after rescue surgery of pelvic recurrence. | After 3 years of median follow-up for living patients.
Overall survival at three years. | After 3 years of median follow-up for living patients.
Disease-free survival at three years | After 3 years of median follow-up for living patients.
Cancer specific survival at three years. | After 3 years of median follow-up for living patients.
Evaluation of anorectal function by using self-administered questionnaire in patients without local recurrence. | 1 year after treatment
Multivariable analysis of prognostic factors associated with clinical complete response. | After 3 years of median follow-up for living patients.

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Bujko, Prof., Principal Investigator — M. Sklodowska-Curie memorial Cancer Centre in Warsaw
Locations (1):
- M. Sklodowska-Curie Memorial Cancer Center, Warsaw, Poland